CLINICAL TRIAL: NCT02815540
Title: The Effects of Cannabidiol (CBD) on Electrical and Autonomic Cardiac Function in Children
Brief Title: The Effects of Cannabidiol (CBD) on Electrical and Autonomic Cardiac Function in Children With Severe Epilepsy
Acronym: CBD1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Investigator no longer at institution, and difficult recruitment; study will not resume
Sponsor: Gillette Children's Specialty Healthcare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CBD-001
Record Dates: First submitted 2016-06-20; First posted 2016-06-28 (Estimated); Results first posted 2022-01-03 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Lennox-Gastaut Syndrome; Dravet Syndrome
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epilepsies, Myoclonic | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Heart Function and Dysautonomia (Other): This study looks at participants already receiving CBD from the state of MN. We are not providing the CBD. We are looking at heart function with ECGs and Holter monitoring before and after CBD is taken by the participant. We are also looking at dysautonomia signs and symptoms and seizure frequency before and after CBD is taken by the participant.
  Interventions: Procedure: 12-Lead ECG; Drug: Cannabidiol

INTERVENTIONS:
Procedure: 12-Lead ECG — Subjects will be monitored while on cannabidiol with a 12-Lead ECG and/or Holter monitoring
  Other Names: Holter Monitor
Drug: Cannabidiol — Subjects who are planning to take state dispensed medical cannabidiol, or are already taking state dispensed medical cannabidiol.

SUMMARY:
The investigators propose to study the effects of cannabidiol (CBD) on cardiac electrical function and the autonomic nervous system in children with Dravet syndrome (DS) and Lennox-Gastaut syndrome (LGS), when the CBD is administered as an artisanal oil obtained through state dispensaries or other sources. The intent is to begin to assess potential risks and benefits of this therapy in a vulnerable patient population by characterizing the effects of CBD on EKG findings, heart rate variability and the occurrence of seizures.

DETAILED DESCRIPTION:
Specific Aims/Study Objectives

This is a pilot study to explore the effects of cannabidiol (CBD) on autonomic cardiac function in children with Dravet syndrome (DS) or Lennox-Gastaut syndrome (LGS) when the CBD is administered as an artisanal oil. This will be achieved by addressing the following specific aims.

Aim #1: To determine the effects of CBD on cardiac function in 30 children with DS and LGS. This is the primary aim of the study: The effects of CBD on the cardiac function of 30 children with DS or LGS will be assessed using a 15-lead electrocardiogram (EKG) and a 24-hour Holter monitor. Investigators hypothesize that there will be no alterations in ventricular repolarization and heart rate variability on the EKG and Holter monitoring, respectively, after taking CBD for 4-8 weeks, compared to when participants were not taking CBD.

Note: The following aims are secondary to the primary outcome and goal of assessing the effects of CBD on cardiac function.

Aim #2: To assess signs and symptoms of dysautonomia in the presence and absence of CBD. Signs and symptoms of dysautonomia include parental perception of body temperature, skin color in hands and feet, sweating, pupil size, flushing, feeding issues, heart rate, strong emotions, constipation, urination or bowel movement issues, and irritability. These signs and symptoms will be collected using a previously-established dysautonomia survey. Investigators hypothesize there will be no change in qualitative assessments of signs and symptoms of dysautonomia after taking CBD for 4-8 weeks, compared to when participants were not taking CBD.

Aim #3: To determine the effects of CBD on the occurrence of seizures. The number of seizures in children who obtain CBD will be assessed using a 7-day seizure diary (Seizure tracker). Caregivers will record the number of seizures for a 7-day period prior to CBD administration, and repeat the seizure tracking after having received CBD for 4-8 weeks. Change in seizure numbers will be compared pre- and post-CBD administration. Investigators hypothesize that study participants will have lower seizure counts after being on CBD compared to when weren't taking CBD.

Study Design and Methodology

Study Design: Thirty patients with DS or LGS who are going to register to take medical cannabis (cannabidiol, or CBD) in the state of Minnesota will be offered the opportunity to participate in this study. If consent is obtained, the patient or guardian will be asked to complete a questionnaire developed for this study that documents observable signs and symptoms of dysautonomia, and to complete a seizure diary for 7 days prior to initially receiving the CBD. Each participant will also have a 15-lead electrocardiogram (EKG) and wear a 24-hour Holter monitor, both non-invasive measures of cardiac function, prior to being administered the CBD. The EKG and 24-hour Holter monitor will be interpreted by a cardiac electrophysiologist and will be reviewed for heart rate variability parameters. The dysautonomia questionnaire, seizure diary and cardiac measurements will be repeated 4-8 weeks after the subject has been on a stable regimen of CBD. This time-frame is based on availability of subjects schedules and clinic visits, and it is also greater than 5 half-lives previously reported for CBD (apparent half-life, 21 hours, (15)). Steady-state levels are achieved after 5 half-lives of drug dosing, thus we expect to be at steady-state concentrations.

Subjects who are already on a stable regimen of CBD, yet plan to stop taking CBD at some point for some reason, are also eligible to participate. The parent or guardian will complete the dysautonomia questionnaire and seizure diary (and research staff will be available to help with questions), and the patient will have the 15-lead EKG and 24-hour Holter monitor while still on the CBD. The subjects will then come back 4-8 weeks after their last dose of CBD to have these assessments repeated while off of the CBD. This time frame is based on availability of subjects schedules and clinic visits as well as being substantially greater than 5 half-lives of CBD, the standard wash-out period for pharmacological studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Dravet syndrome or Lennox-Gastaut syndrome
* Patients who are planning to obtain medical cannabidiol
* Patients who are already taking medical cannabidiol and are planning to stop taking it

Exclusion Criteria:

* Patients without a diagnosis of Dravet syndrome or Lennox-Gastaut syndrome

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly S Wical, MD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Dravet C, Bureau M, Oguni H, Fukuyama Y, Cokar O. Severe myoclonic epilepsy in infancy (Dravet syndrome). In: Roger J, Bureau M, Dravet C, Genton P, Tassinari CA, Wolf P (eds) Epileptic syndromes in infancy, childhood and adolescence, 4th ed. John Libbey, London, 2005, pp 89 - 109.
- [Background] 2. http://www.ninds.nih.gov/disorders/lennoxgastautsyndrome/lennoxgastautsyndrome.htm, Retrieved 6.10.2015
- [Background] Sakauchi M, Oguni H, Kato I, Osawa M, Hirose S, Kaneko S, Takahashi Y, Takayama R, Fujiwara T. Mortality in Dravet syndrome: search for risk factors in Japanese patients. Epilepsia. 2011 Apr;52 Suppl 2:50-4. doi: 10.1111/j.1528-1167.2011.03002.x. PMID 21463280
- [Background] Skluzacek JV, Watts KP, Parsy O, Wical B, Camfield P. Dravet syndrome and parent associations: the IDEA League experience with comorbid conditions, mortality, management, adaptation, and grief. Epilepsia. 2011 Apr;52 Suppl 2:95-101. doi: 10.1111/j.1528-1167.2011.03012.x. PMID 21463290
- [Background] Jehi L. Sudden death in epilepsy, surgery, and seizure outcomes: the interface between heart and brain. Cleve Clin J Med. 2010 Jul;77 Suppl 3:S51-5. doi: 10.3949/ccjm.77.s3.09. PMID 20622077
- [Background] Kalume F. Sudden unexpected death in Dravet syndrome: respiratory and other physiological dysfunctions. Respir Physiol Neurobiol. 2013 Nov 1;189(2):324-8. doi: 10.1016/j.resp.2013.06.026. Epub 2013 Jul 9. PMID 23850567
- [Background] 7. Wical, B, Wendorf H, Leighty D, Tervo M, Tervo R. Signs of Dysautonomia in Children with Dravet Syndrome. Presented at the Annual Meeting of the American Epilepsy Society, Boston, MA, Dec 2009.
- [Background] Delogu AB, Spinelli A, Battaglia D, Dravet C, De Nisco A, Saracino A, Romagnoli C, Lanza GA, Crea F. Electrical and autonomic cardiac function in patients with Dravet syndrome. Epilepsia. 2011 Apr;52 Suppl 2:55-8. doi: 10.1111/j.1528-1167.2011.03003.x. PMID 21463281
- [Background] Nei M, Sperling MR, Mintzer S, Ho RT. Long-term cardiac rhythm and repolarization abnormalities in refractory focal and generalized epilepsy. Epilepsia. 2012 Aug;53(8):e137-40. doi: 10.1111/j.1528-1167.2012.03561.x. Epub 2012 Jun 18. PMID 22709423
- [Background] Ergul Y, Ekici B, Tatli B, Nisli K, Ozmen M. QT and P wave dispersion and heart rate variability in patients with Dravet syndrome. Acta Neurol Belg. 2013 Jun;113(2):161-6. doi: 10.1007/s13760-012-0140-z. Epub 2012 Oct 13. PMID 23065439
- [Background] Granjeiro EM, Gomes FV, Guimaraes FS, Correa FM, Resstel LB. Effects of intracisternal administration of cannabidiol on the cardiovascular and behavioral responses to acute restraint stress. Pharmacol Biochem Behav. 2011 Oct;99(4):743-8. doi: 10.1016/j.pbb.2011.06.027. Epub 2011 Jul 12. PMID 21771609
- [Background] Bergamaschi MM, Queiroz RH, Chagas MH, de Oliveira DC, De Martinis BS, Kapczinski F, Quevedo J, Roesler R, Schroder N, Nardi AE, Martin-Santos R, Hallak JE, Zuardi AW, Crippa JA. Cannabidiol reduces the anxiety induced by simulated public speaking in treatment-naive social phobia patients. Neuropsychopharmacology. 2011 May;36(6):1219-26. doi: 10.1038/npp.2011.6. Epub 2011 Feb 9. PMID 21307846
- [Background] Martin-Santos R, Crippa JA, Batalla A, Bhattacharyya S, Atakan Z, Borgwardt S, Allen P, Seal M, Langohr K, Farre M, Zuardi AW, McGuire PK. Acute effects of a single, oral dose of d9-tetrahydrocannabinol (THC) and cannabidiol (CBD) administration in healthy volunteers. Curr Pharm Des. 2012;18(32):4966-79. doi: 10.2174/138161212802884780. PMID 22716148
- [Background] Gloss D, Vickrey B. Cannabinoids for epilepsy. Cochrane Database Syst Rev. 2014 Mar 5;2014(3):CD009270. doi: 10.1002/14651858.CD009270.pub3. PMID 24595491
- [Background] 15. Ohlsson A, Lindgren JE, Andersson S, Agurell S, Gillespie H, Hollister L. (1984). Single dose kinetics of cannabidiol in man. Cannabinoids: chemical, pharmacologic, and therapeutic aspects. S. Agurell, W. L. Dewey and R. Willette. Orlando, FL, Academic Press Inc.: 219-225. doi: 10.1016/B978-0-12-044620-9.50003-8

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Heart Function and Dysautonomia
Started | 2
Completed | 0
Not Completed | 2
Not completed — Physician left institution and study was discontinued. No other PI was available. | 2

BASELINE CHARACTERISTICS:
Groups:
- Observational: This study looks at participants already receiving CBD from the state of MN. We are not providing the CBD. We are looking at heart function with ECGs and Holter monitoring before and after CBD is taken by the participant. We are also looking at dysautonomia signs and symptoms and seizure frequency before and after CBD is taken by the participant.
  12-Lead ECG: Subjects will be monitored while on cannabidiol with a 12-Lead ECG and/or Holter monitoring
  Cannabidiol: Subjects who are planning to take state dispensed medical cannabidiol, or are already taking state dispensed medical cannabidiol.
Arm/Group | Observational
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Holter SDNN Parameter Change
Description: Change from baseline Holter SDNN parameter to follow up visit Holter SDNN parameter.
Time Frame: Baseline to 4 to 8 week follow up visit
Population: Physician left institution and study was discontinued due to no other investigators available.
Arm/Group | Heart Function and Dysautonomia
Number analyzed (Participants) | 0

2. Secondary Outcome: Seizure Frequency
Description: Change from baseline seizure frequency to follow up visit seizure frequency.
Time Frame: Baseline and 4 to 8 week follow up visit
Population: Physician left institution and study was discontinued due to no other investigators available.
Arm/Group | Heart Function and Dysautonomia
Number analyzed (Participants) | 0

3. Secondary Outcome: Dysautonomia Signs and Symptoms
Description: signs and symptoms assessed by questionnaire developed for this study that documents observable signs and symptoms of dysautonomia
Time Frame: Baseline and 4 to 8 week follow up visit
Population: Physician left institution and study was discontinued due to no other investigators available.
Arm/Group | Heart Function and Dysautonomia
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: No data were collected.
Description: No data were collected.
Arm/Group | Observational
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Physician left institution and study was discontinued due to no other investigators available. No outcome measures were collected or analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT02815540/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT02815540/ICF_001.pdf